CLINICAL TRIAL: NCT06107322
Title: Retrospective Study on the Hematological Effects of Atypical Antipsychotics (AAPs) in a Geriatric Population: What is the Role of 5-HT2 Receptors
Brief Title: Hematological Effects of Atypical Antipsychotics (AAPs) in a Geriatric Population: What is the Role of 5-HT2 Receptors
Acronym: AAPs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8902
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Neutropenia
Keywords: Neutropenia; Atypical antipsychotics (AAPs); 5-HT2 receptors; Hematological effects
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
White lineage abnormalities and in particular neutropenia and agranulocytosis are known and increasingly studied adverse effects of antipsychotics, particularly second generation. White lineage abnormalities have been found with each of the drugs in this class even if progression to agranulocytosis is rarer with drugs other than Clozapine.

The infections, sometimes serious, induced by these adverse effects have largely led to limiting the use of second generation antipsychotics, and in particular clozapine, to the treatment of patients resistant to other first or second line treatments.

Several hypotheses have been put forward: the first is that of an immuno-allergic reaction mediated by eosinophils with increased sensitivity depending on the HLA type, another that of a direct toxic effect of clozapine or its main metabolite, N -demethylclozapine and a third attributes hematological disorders to catecholaminergic inhibition which prevents the differentiation of CD34+ hematopoietic stem cells into leukocytes, after blocking dopaminergic and/or beta-adrenergic receptors.

More recently, a new hypothesis is emerging following scandals particularly in France linked to Benfluorex (Mediator®), Dexfenfluramine (Isomeride®) and Fenfluramine (Pondéral®). Indeed, by studying the cellular mechanisms linked to the stimulation of the 5-HT2B receptor by their common metabolite Nordexfenfluramine, researchers from the NeuroCardiovascular pharmacology and toxicology laboratory in Strasbourg have demonstrated that the stimulation of 5-HT2BR mobilizes CD34+ cells in blood from the bone marrow and selective blocking of 5-HT2B receptors, reduces the number of leukocytes in the blood, mainly neutrophils and lymphocytes, further decreasing their blood concentration with exposure time.

DETAILED DESCRIPTION:
The investigators chose as their study population an elderly to very elderly population, hospitalized or residing in the Geriatrics center of a university hospital. Indeed, apart from resistant schizophrenia, clozapine is the reference antipsychotic in behavioral disorders associated with the dementia of Parkinson's disease, Lewy body disease and other atypical parkinsonian syndromes, particularly because of its antagonism. dopaminergic less important. The absence of equivalent therapy justifies studying the occurrence of adverse effects precisely in this population. Studies have already taken place on clozapine in this indication but to our knowledge none have sought to demonstrate the occurrence of white lineage disorders based on its effects on 5-HT2 receptors.

This study could provide a better understanding of the role and function of serotonin receptors of the 5-HT2 subtype, on the differentiation/mobilization of hematopoietic cells, with the clinical challenge of better prescription in the geriatric population, often fragile, of atypical neuroleptics which are the only therapeutic alternative in the delusional disorders of patients with Lewy bodies but also used in other neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 65 years old)
* Subject hospitalized in Geriatric Internal Medicine, in Geriatric Follow-up Care and Rehabilitation, in a Long-Term Care Unit or Important Medical-Technical Care, in a Reinforced Accommodation Unit or in a Cognitive-Behavioral Unit at Strasbourg University Hospitals)
* Subject not opposing the reuse of their data for the purposes of this research.
* Indication for the introduction of the neuroleptic indicated
* Available dosage and frequency of administration and duration of treatment

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Presence of a neuroleptic before admission to the University Hospitals of Strasbourg, excluding readmission of a patient included
* Neuroleptics not present on the discharge prescription for long-term treatment
* Neuroleptics prescribed for less than 48 hours
* Presence of a white lineage anomaly prior to the initiation of neuroleptic treatment
* Patient contraindicated for taking a long-term neuroleptic.
* Hematological disease with white lineage abnormality (lymphoma, leukemia, myelodysplasia, mye syndrome

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Major subject (≥ 65 years old) having indication for the introduction of the neuroleptic indicated
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-23 (Estimated)

PRIMARY OUTCOMES:
Number of neutrophils per liter of blood | 1 hour after blood collection

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pharmacie - Stérilisation - CHU de Strasbourg - France, Strasbourg, France